CLINICAL TRIAL: NCT00922415
Title: Use of Fecal Calprotectin as a Surrogate Marker for Macroscopic Recurrence of Disease in Patients With Crohn's Disease After Intestinal Resection
Brief Title: Fecal Calprotectin as a Marker for Macroscopic Recurrence of Crohn's Disease After Intestinal Resection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Dr. Iris Dotan, Dep. of Gastroenterology, Tel Aviv medical center
Other Study IDs: TASMC-09-ID-255-CTIL; 255-09
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-12

CONDITIONS: Complicated Crohn's Disease
Keywords: Crohn's disease; calprotectin
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — At all follow-up visits, they will undergo the following tests; CBC, ESR, CRP, and fecal calprotectin. Sera will be stored for antibodies such as ASCA or anti glycan antibodies.
  During colonoscopy, disease recurrence will be evaluated by two scores, the Rutgeerts score and the CDEIS score, both containing 4 grades. Recurrence will be assessed by histological findings as well.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cases: patients at least 18 years of age, with confirmed Crohn's disease undergoing intestinal resection for complicated Crohn's disease

SUMMARY:
our primary objective is to correlate fecal calprotectin with currently used Crohn's disease endoscopic disease activity scores used for predicting endoscopic recurrence. Our secondary objectives will be to determine a cutoff for early macroscopic recurrence of disease based on surveillance colonoscopies , and to compare this with other surrogate markers .

DETAILED DESCRIPTION:
Fecal calprotectin is a non invasive marker of intestinal inflammation. It is highly sensitive for the detection of active Crohn's disease (13) and mucosal healing (14). Levels higher than 250 mg/L are associated with relapse, and levels < 50 usually with remission. Mucosal healing was noted in patients with calprotectin levels less < 130 mg/L, and a mean level < 30 mg/L (13,14) .It is therefore an excellent candidate for a simple clinically available surrogate marker for endoscopic recurrence after intestinal resection in Crohn's disease. In the current study, our primary objective is to correlate fecal calprotectin with currently used Crohn's disease endoscopic disease activity scores used for predicting endoscopic recurrence. Our secondary objectives will be to determine a cutoff for early macroscopic recurrence of disease based on surveillance colonoscopies , and to compare this with other surrogate markers .

Methods This will be a prospective non-interventional observational study, performed at the Sourasky Medical center in Tel Aviv, over two years.

Patients with confirmed Crohn's disease undergoing intestinal resection for complicated Crohn's disease - will be followed for one year, and undergo a follow- up colonoscopy between 6-9 months after surgery. Patients will be seen at enrollment and follow-up visits, 3,6,9& 12 months after surgery. At enrollment, sites of disease, age of onset, smoking history and previous medication use will be registered, as well as presence of strictures and fistula, or previous surgery. At all visits, patients will be questioned regarding disease symptoms, smoking, and medication use. During each of the follow-up visits, patients will be examined, weighed, and have a disease activity index recorded. At all follow-up visits, they will undergo the following tests; CBC, ESR, CRP, and fecal calprotectin. Sera will be stored for antibodies such as ASCA or anti glycan antibodies.

During colonoscopy, disease recurrence will be evaluated by two scores, the Rutgeerts score and the CDEIS score, both containing 4 grades. Recurrence will be assessed by histological findings as well.

End points For the primary outcome, we will check if calprotecin levels are correlated with endoscopic scores. We will also evaluate cutoffs of calprotectin that are correlated with grade 3 or 4 Rutgeerts or CDEIS.

Other secondary endpoints will include:

Correlation between calprotectin and early clinical relapse (within one year) Correlation between calprotectin and histologic relapse (within one year) Correlation between anti glycan antibodies and early clinical relapse (within one year) Correlation between CDEIS and antiglycan antibodies

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* confirmed Crohn's disease
* undergoing intestinal resection for complicated Crohn's disease

Exclusion Criteria:

* Ileostomy
* pregnancy
* stricturoplasty without resection
* patients with diffuse active disease at other sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients at least 18 years of age, with confirmed Crohn's disease undergoing intestinal resection for complicated Crohn's disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-08 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
we will check if calprotectin levels are correlated with endoscopic scores and with grade 3 or 4 Rutgeerts or CDEIS. | once, at colonoscopy

SECONDARY OUTCOMES:
Correlation between calprotectin and early clinical relapse | within one year
Correlation between calprotectin and histologic relapse | within one year
Correlation between anti glycan antibodies and early clinical relapse | within one year
Correlation between CDEIS and antiglycan antibodies | at colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Dep. of Gastroenterology, Tel Aviv medical center, Tel Aviv, Israel